CLINICAL TRIAL: NCT02270996
Title: An Antimicrobial Stewardship Intervention Program in Pediatric Surgery
Brief Title: Antimicrobial Stewardship in Pediatric Surgery
Acronym: AbxPS
Status: Withdrawn | Type: Observational
Sponsor: Alberta Children's Hospital (Other)
Responsible Party: Principal Investigator, Dr Anna Shawyer, Dr. Anna Shawyer, Alberta Children's Hospital
Other Study IDs: ACH PedSurg ACS 002
Record Dates: First submitted 2014-10-08; First posted 2014-10-22 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Appendicitis
Keywords: antibiotic, antimicrobial, stewardship, child
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NO Antimicrobial Stewardship Program: Prospective cohort of children who undergo appendectomy for acute appendicitis (perforated and non-perforated) BEFORE the implementation of the Antimicrobial Stewardship Program.
- WITH Antimicrobial Stewardship Program: Prospective cohort of children who undergo appendectomy for acute appendicitis (perforated and non-perforated) WITH the implementation of the Antimicrobial Stewardship Program.
  Interventions: Other: Antimicrobial Stewardship Program

INTERVENTIONS:
Other: Antimicrobial Stewardship Program — Twice weekly meeting with Infectious Disease and Pediatric Surgery team members to audit antibiotics prescribed and suggest role for discontinuation.
  Groups: WITH Antimicrobial Stewardship Program

SUMMARY:
Acute appendicitis is a common surgical emergency in children. Non-perforated appendicitis patients do not require antibiotics after appendectomy. Although guidelines and recommendations exist to decrease post-operative antibiotic mis-use after appendectomy, surgeons continue to prescribe unwarranted antibiotics.

The aim of this study is to determine if an Antimicrobial Stewardship Program in Pediatric Surgery will decrease the use of un-warranted antibiotics.

DETAILED DESCRIPTION:
Many surgeons continue to treat non-perforated or "borderline perforated" appendicitis with postoperative antibiotics despite an evidence-based definition of perforation (in the pediatric surgical literature) and many guidelines and recommendations that specify that no postoperative antibiotics are required. Children with perforated appendicitis are also often treated with longer-than-necessary courses of antibiotics. Although surgeons may feel that they only prescribe additional doses on occasion, evidence suggests that this behavior occurs in over 50% of children with non-perforated appendicitis.

These additional doses contribute to a longer length of stay, excess costs to the health care system, and disrupt patient flow. Additionally, the patients are exposed to more antibiotics and their potential for adverse effects (such as incorrect dose, incorrect medication, allergic reaction, antimicrobial resistance or c difficile infection).

Antimicrobial stewardship programs have been successful in pediatrics and adult general surgery in curbing unwarranted antibiotic use, but have never been evaluated in pediatric general surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participant (surgeon) is a pediatric surgeon at McMaster Children's Hospital and takes care of patients under the age of 18 who undergo appendectomy.
* Participant (surgeon) is able to read, write and understand English.
* Participant (surgeon) is able to provide informed consent.

Exclusion Criteria:

* Participant (surgeon) only has patients who undergo drain insertion, PICC line insertion or a secondary operation during the same admission
* Participant (surgeon) only has patients who do not undergo operation (i.e. "conservative management with interval appendectomy)
* Participant (surgeon) does not provide informed consent
* Participant (surgeon) does not understand written and spoken English diagnosis other than appendicitis at time of operation

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population is the pediatric surgeons at our institution who will have their antibiotic prescribing audited.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Compliance with American Pediatric Surgical Association recommendations for postoperative antibiotics for appendicitis | From date of admission until first follow-up visit, typically within 4-6 weeks of discharge
  Includes both intravenous and oral antibiotics prescribed, both during the time frame from admission until discharge, in addition to any prescription given for home, oral antibiotics. Measured as yes/no

SECONDARY OUTCOMES:
Postoperative intravenous antibiotics for non-perforated appendicitis | From date of admission until first follow-up visit, typically within 4-6 weeks of discharge
  measured as number of days (ie number of doses divided by number of doses-per-day)
Postoperative oral antibiotics for non-perforated appendicitis | From date of admission until first follow-up visit, typically within 4-6 weeks of discharge
  measured as number of days (ie number of doses divided by number of doses-per-day)

OTHER OUTCOMES:
Postoperative fever | Length of admission
  Rectal temperature above 100.4ºF (38ºC), measured as yes/no and on what postoperative day Oral temperature above 100ºF (37.8ºC) Axillary (armpit) temperature above 99ºF (37.2ºC) Ear (tympanic membrane) temperature above 100.4ºF (38ºC) in rectal mode or 99.5ºF (37.5ºC) in oral mode Forehead (temporal artery) temperature above 100.4ºF (38ºC)
Readmission within 30 days | Within 30 days of discharge
  Need for readmission within 30 days of discharge, measured as yes/no
Peripherally inserted intravenous catheter (PICC) | From date of admission until first follow-up visit, typically within 4-6 weeks of discharge
  Need for PICC insertion for long term antibiotics, intravenous fluids or parenteral nutrition, measured as yes/no
Drain insertion | From date of admission until first follow-up visit, typically within 4-6 weeks of discharge
  Need for a drain insertion (by interventional radiology) for postoperative abscess, measured as yes/no
Re-operation | From date of admission until first follow-up visit, typically within 4-6 weeks of discharge
  Need for re-operation on the same admission, measured as yes/no
Length of Stay | Length of admission
  Measured in days (from date of admission until date of discharge)
Adverse reaction to antibiotic | From date of admission until first follow-up visit, typically within 4-6 weeks of discharge
  Measured as yes/no in addition to description of reaction (eg hives, shortness of breath)
Wrong medication/Wrong dose | From date of admission until date of first follow-up visit, typically within 4-6 weeks of discharge
  Measured as yes/no in addition to description of problem (wrong dose, wrong medication)
C difficile infection | From date of admission until first follow-up visit, typically within 4-6 weeks of discharge
  Measured as yes/no based on stool assay

CONTACTS AND LOCATIONS:
Overall Officials: Anna Shawyer, MS, MSc, Principal Investigator — Alberta Children's Hospital

REFERENCES:
- [Result] St Peter SD, Sharp SW, Holcomb GW 3rd, Ostlie DJ. An evidence-based definition for perforated appendicitis derived from a prospective randomized trial. J Pediatr Surg. 2008 Dec;43(12):2242-5. doi: 10.1016/j.jpedsurg.2008.08.051. PMID 19040944
- [Result] Lee SL, Islam S, Cassidy LD, Abdullah F, Arca MJ; 2010 American Pediatric Surgical Association Outcomes and Clinical Trials Committee. Antibiotics and appendicitis in the pediatric population: an American Pediatric Surgical Association Outcomes and Clinical Trials Committee systematic review. J Pediatr Surg. 2010 Nov;45(11):2181-5. doi: 10.1016/j.jpedsurg.2010.06.038. PMID 21034941
- [Result] Srigley JA, Brooks A, Sung M, Yamamura D, Haider S, Mertz D. Inappropriate use of antibiotics and Clostridium difficile infection. Am J Infect Control. 2013 Nov;41(11):1116-8. doi: 10.1016/j.ajic.2013.04.017. Epub 2013 Aug 7. PMID 23932828
- [Result] Rangel SJ, Fung M, Graham DA, Ma L, Nelson CP, Sandora TJ. Recent trends in the use of antibiotic prophylaxis in pediatric surgery. J Pediatr Surg. 2011 Feb;46(2):366-71. doi: 10.1016/j.jpedsurg.2010.11.016. PMID 21292089
- [Result] Ghaleb MA, Barber N, Franklin BD, Wong IC. The incidence and nature of prescribing and medication administration errors in paediatric inpatients. Arch Dis Child. 2010 Feb;95(2):113-8. doi: 10.1136/adc.2009.158485. Epub 2010 Feb 4. PMID 20133327